CLINICAL TRIAL: NCT00847886
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose Study to Determine the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of LX3305 and Methotrexate in Subjects With Stable Rheumatoid Arthritis
Brief Title: Study of LX3305 and Methotrexate in Subjects With Stable Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Joel P. Freiman, MD, MPH (Medical Director, Drug Safety), Lexicon Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Protocol LX3305.1-104-DDI; LX3305.104; LX2931
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Results first posted 2010-06-03 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LX3305 (Experimental): Daily oral intake of LX3305 for 14 days.
  Interventions: Drug: LX3305; Drug: Methotrexate
- LX3305 Placebo (Placebo Comparator): Matching placebo dosing with daily oral intake for 14 days.
  Interventions: Drug: LX3305 Placebo; Drug: Methotrexate

INTERVENTIONS:
Drug: LX3305 — Daily oral intake of LX3305 for 14 days.
  Arms: LX3305
Drug: LX3305 Placebo — Matching placebo dosing with daily oral intake for 14 days.
  Arms: LX3305 Placebo
Drug: Methotrexate — Once weekly stable-dose methotrexate.

SUMMARY:
The purpose of the study is to evaluate the effect of LX3305 on methotrexate (MTX) pharmacokinetics and to evaluate the safety and tolerability of LX3305 given over 14 days in subjects with stable rheumatoid arthritis that are receiving stable doses of MTX.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years old
* Must be willing to practice 2 adequate methods of contraception for the duration of the study
* Rheumatoid arthritis present for at least 3 months; functional class I, II, or III as defined by ACR criteria
* Treatment with methotrexate (7.5 to 25 mg per week) for at least the last 3 months, and currently receiving stable dose methotrexate for at least one month prior to the start of the study
* Ability to provide written informed consent

Exclusion Criteria:

* Women who are pregnant or nursing
* History of other current inflammatory arthritis
* History of opportunistic infection
* History of recurrent infections or current infection 2 weeks prior to start of study
* Presence of significant, uncontrolled medical problems
* Treatment with any disease-modifying anti-rheumatoid drugs other than methotrexate within 4 weeks prior to start of study
* Use of chondroitin sulfate, glucosamine sulfate, minocycline, or matrix metalloproteinase inhibitors, H-2 blockers, proton pump inhibitors, or misoprostol within 4 weeks prior to study start
* Receipt of live vaccine within 8 weeks prior to study start
* Rheumatoid arthritis, functional class IV as defined by ACR criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip M. Brown, MD, JD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (1):
- Metroplex Clinical Research Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was performed at one center in Dallas, TX. Recruitment began in January 2009 and the last subject completed the study in March 2009.
Pre-assignment Details: One subject did not complete the study due to an adverse event of uveitis on Day 1 and was not dosed with study drug. This subject was not included in any population analyses. Therefore, the participant flow includes 15 subjects, 12 receiving active drug and 3 receiving placebo.
Groups:
- LX3305 + Methotrexate: Daily oral intake of 100 mg LX3305 for 14 days.
- Methotrexate: Matching placebo dosing with daily oral intake for 14 days.
Period: Overall Study
Arm/Group | LX3305 + Methotrexate | Methotrexate
Started | 12 | 4
Completed | 12 | 3
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LX3305 + Methotrexate | Methotrexate | Total
Number analyzed (Participants) | 12 | 3 | 15
Age Continuous [Mean (Standard Deviation); unit: years] | 59.8 (10.25) | 58.7 (14.74) | 59.5 (10.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 3 | 15
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Methotrexate Maximum Plasma Concentration
Time Frame: Day 15
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LX3305 + Methotrexate | Methotrexate
Number analyzed (Participants) | 12 | 3
ng/mL | 215 (71.4) | 177 (72.1)

2. Primary Outcome: Time to Reach Maximum Plasma Concentration of Methotrexate
Time Frame: Day 15
Measure: Median (Full Range); unit: hours
Arm/Group | LX3305 + Methotrexate | Methotrexate
Number analyzed (Participants) | 12 | 3
hours | 0.98 [0.90 to 2.98] | 1.25 [1.00 to 3.00]

3. Primary Outcome: Half-life of Methotrexate in Plasma
Time Frame: Day 15
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | LX3305 + Methotrexate | Methotrexate
Number analyzed (Participants) | 12 | 3
hours | 3.80 (0.520) | 3.80 (0.693)

4. Primary Outcome: Amount of Methotrexate Excreted in the Urine
Time Frame: Day 15
Measure: Mean (Standard Deviation); unit: µg
Arm/Group | LX3305 + Methotrexate | Methotrexate
Number analyzed (Participants) | 12 | 3
µg | 3861 (1720) | 4022 (1218)

5. Primary Outcome: 7-Hydroxymethotrexate (7-OH-MTX) Maximum Plasma Concentration
Description: 7-OH-MTX is the primary metabolite of methotrexate.
Time Frame: Day 15
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LX3305 + Methotrexate | Methotrexate
Number analyzed (Participants) | 12 | 3
ng/mL | 25.5 (12.8) | 25.5 (15.4)

6. Primary Outcome: Time to Reach Maximum Plasma Concentration of 7-OH-MTX
Time Frame: Day 15
Measure: Median (Full Range); unit: hours
Arm/Group | LX3305 + Methotrexate | Methotrexate
Number analyzed (Participants) | 12 | 3
hours | 6.01 [5.90 to 11.98] | 8.00 [4.00 to 12.00]

7. Primary Outcome: Amount of 7-OH-MTX Excreted in the Urine
Time Frame: Day 15
Measure: Mean (Standard Deviation); unit: µg
Arm/Group | LX3305 + Methotrexate | Methotrexate
Number analyzed (Participants) | 12 | 3
µg | 285 (106) | 281 (109)

8. Secondary Outcome: Maximum Plasma Concentration of LX3305 in the Presence of MTX
Time Frame: Day 15
Population: This outcome was not measured in the Methotrexate + LX3305 placebo subjects.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LX3305 + Methotrexate | Methotrexate
Number analyzed (Participants) | 12 | 0
ng/mL | 588 (233) |

9. Secondary Outcome: Time to Maximum Plasma Concentration of LX3305 in the Presence of MTX
Time Frame: Day 15
Population: This outcome was not measured in the Methotrexate + LX3305 placebo subjects.
Measure: Median (Full Range); unit: hours
Arm/Group | LX3305 + Methotrexate | Methotrexate
Number analyzed (Participants) | 12 | 0
hours | 2.25 [1.42 to 4.00] |

10. Secondary Outcome: Half-life of LX3305 in Plasma in the Presence of MTX
Time Frame: Day 15
Population: This outcome was not measured in the Methotrexate + LX3305 placebo subjects.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | LX3305 + Methotrexate | Methotrexate
Number analyzed (Participants) | 12 | 0
hours | 5.89 (1.54) |

11. Secondary Outcome: Percentage of Change From Baseline in Absolute Total Lymphocyte Count at Day 15
Description: Baseline was defined as pre-dose on Day 1.
Time Frame: Day 15
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | LX3305 + Methotrexate | Methotrexate
Number analyzed (Participants) | 12 | 3
Percent | -14.049 (29.1505) | -6.152 (15.0143)

ADVERSE EVENTS:
Time Frame: 22 days
Description: An adverse event is defined as any noxious, pathological, or unintended change in anatomical, physiological, or metabolic functions as indicated by physical signs or symptoms occurring in any phase of the clinical study whether or not associated with the study medication and whether or not considered related to the study medication.
Arm/Group | LX3305 + Methotrexate | Methotrexate
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/3
Other Adverse Events (participants affected / at risk) | 10/12 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LX3305 + Methotrexate (N=12) | Methotrexate (N=3)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea hemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 1 (1)
Athralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Eye swelling (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperemia (Eye disorders) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor requires that written permission be given before the investigator can release any data publicly.